CLINICAL TRIAL: NCT04649138
Title: Fomepizole Dosing During Continuous Renal Replacement Therapy (CRRT)
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, Knut Erik Hovda, MD, PhD, Principal Investigator, Oslo University Hospital
Other Study IDs: 2017/981
Record Dates: First submitted 2020-10-30; First posted 2020-12-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2020-11

CONDITIONS: Toxic Alcohol Poisoning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The project is a prospective observation study of patients with suspected or confirmed toxic alcohol poisoning treated with fomepizole and continuous renal replacement therapy (CRRT)

ELIGIBILITY:
Inclusion Criteria:

* Patients (over 18 year) with suspected or confirmed toxic alcohol poisoning treated with fomepizole and CRRT.

Exclusion Criteria:

* Patients who wish to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Toxic alcohol poisoning treated with fomepizole and CRRT.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Measure minimum plasma concentration of fomepizole | through study completion, up to 72 hours
  Plasma samples will be obtained up to every hour and before fomepizole is given

SECONDARY OUTCOMES:
Continuous renal replacement therapy (CRRT) clearance of fomepizole | through study completion, up to 72 hours
  Plasma and dialysat samples will be obtained up to every hour
Determine saturation/sieving coefficient of fomepizole | through study completion, up to 72 hours
  Plasma and dialysat samples will be obtained up to every hour

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No